CLINICAL TRIAL: NCT07156006
Title: Automatic Quantification of Breast Arterial Calcifications as an Imaging Biomarker of Cardiovascular Risk (the BAKER Study)
Brief Title: Breast Arterial Calcifications as an Imaging Biomarker of Cardiovascular Risk
Acronym: BAKER
Status: Terminated | Type: Observational
Why Stopped: PI ceased activity
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Francesco Sardanelli, Director, IRCCS Policlinico S. Donato
Other Study IDs: BAKER; 90/INT/2020 (Other: Comitato Etico Territoriale Lombardia 1)
Record Dates: First submitted 2024-01-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Breast; Cardiovascular Calcification
MeSH Terms: interventions — Mammography; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- BAC Group: Outpatients presenting in our department for annual mammography will be screened and selected for BAC presence.
  Mammographic Imaging:
  Participants will undergo mammographic imaging using a digital full-field mammography system, following standard clinical practices.
  The acquired mammographic images will serve as the basis for the development and testing of the Convolutional Neural Network (CNN) for Breast Arterial Calcifications (BAC) segmentation.
  Venous Blood Sample Collection:
  For each participants, a venous blood sample will be collected and traditional cardiovascular risk factors (such as age, hypertension, hyperlipidemia) will be recorded.
  Interventions: Diagnostic Test: Mammography
- Control Group: Outpatients presenting in our department for annual mammography will be screened and matched for age and breast density to BAC Group.
  Mammographic Imaging:
  Participants will undergo mammographic imaging using a digital full-field mammography system, following standard clinical practices.
  The acquired mammographic images will serve as the basis for the development and testing of the Convolutional Neural Network (CNN) for Breast Arterial Calcifications (BAC) segmentation.
  Venous Blood Sample Collection:
  For each participants, a venous blood sample will be collected and traditional cardiovascular risk factors (such as age, hypertension, hyperlipidemia) will be recorded.
  Interventions: Diagnostic Test: Mammography

INTERVENTIONS:
Diagnostic Test: Mammography — Participants will undergo mammographic imaging using a digital full-field mammography system, following standard clinical practices and blood sampling.
  Other Names: Blood test

SUMMARY:
The goal of this observational study is to assess if there is an association between the presence of BAC and traditional cardiovascular risk factors and validate a Convolutional Neural Network (CNN) for the automatic segmentation of Breast Arterial Calcifications (BAC) in mammographic images. This study focuses on understanding the potential of BAC as an imaging biomarker for cardiovascular risk.

The main questions it aims to answer are:

* Is there an association between the presence of BAC and traditional cardiovascular risk factors?
* Can a CNN accurately segment BAC in mammographic images?
* What is the correlation between BAC and White Matter Hyperintensities (WMH) detected through brain MRI?

Participants in this study will be individuals who undergo mammographic screening. The main tasks participants will be asked to do include providing consent for participation and having mammographic images and a blood sample taken. The study will use a comparison group, comparing individuals with BAC to those without BAC, to assess potential effects on cardiovascular risk.

DETAILED DESCRIPTION:
Association between BAC and Cardiovascular Risk Factors

* Traditional cardiovascular risk factors will be analyzed, and statistical tests (t-test or U de Mann-Whitney) will be employed based on the data distribution.
* Multivariate analysis will be performed to determine the independent association between BAC load and cardiovascular risk factors.
* Linear regression will assess the relationship between BAC load and Framingham score, aiming for a clinically applicable model.

Development of CNN for BAC Segmentation

* Mammographic images will be acquired using a digital full-field mammography system as per clinical practice.
* Two experienced operators will manually segment the images to create a dataset for training, validation, and testing the CNN.
* About 60% of the images acquired in the first year will be used for training, and the remaining 40% will form the validation and test datasets.
* Performance evaluation of the CNN will be conducted using the Sørensen similarity index, Bland-Altman analysis, and Free Response Receiver Operating Characteristic (FROC).

Association between BAC and White Matter Hyperintensities (WMH)

* A subset of participants will undergo brain MRI to assess WMH.
* The association between BAC quantity in mammography and WMH load in MRI will be evaluated using machine learning techniques.
* Other small vessel disease markers, such as lacunar infarcts and microbleeds, will also be analyzed.

Patient Enrollment:

The study aims to enroll 600 women, considering a 1:1 ratio between cases and controls. With an estimated 50% adherence rate, it anticipates evaluating 1500 women over two years.

This comprehensive study integrates the development of advanced imaging techniques with clinical correlations to explore the potential of BAC as an imaging biomarker for cardiovascular risk assessment.

ELIGIBILITY:
Inclusion Criteria:

Female participants. Consent to undergo mammography screening. Agreement to participate in brain MRI for a subset of the study.

Exclusion Criteria:

Male participants. Age below 40. Inability or unwillingness to undergo mammography screening. Contraindications for brain MRI, including the presence of pacemaker, intracranial ferromagnetic vascular clips, intraocular metallic fragments, severe claustrophobia, inability to maintain a supine position, involuntary movements, or pregnancy.

Known history of breast cancer. Previous reductive breast surgery.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of women aged more than 40 years who have consented to undergo mammography screening. Participants will be recruited from individuals attending mammography screening programs at our institute.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Association Between BAC and Cardiovascular Risk Factors | One observation at the time of the mammography examination. Total time frame: 1 day.
  Methodology: This aspect of the study aims to assess the association between the burden of BAC and traditional cardiovascular risk factors. Parametric and non-parametric tests will be employed to evaluate differences in BAC burden based on the presence or absence of traditional cardiovascular and gynecological risk factors.
  Implications: A positive association between BAC burden and cardiovascular risk factors may emphasize the potential of BAC as a biomarker for cardiovascular risk.

SECONDARY OUTCOMES:
Diagnostic Performance of CNN Detection and Quantification of BAC on Mammograms | One observation at the time of the mammography examination. Total time frame: 1 day.
  To assess the performance and accuracy of the Convolutional Neural Network (CNN) in automatically segmenting BAC from mammographic images. The assessment will be based on metrics such as the Sørensen similarity index, Bland-Altman analysis, and Free Response Receiver Operating Characteristic (FROC) analysis. The CNN's ability to reliably and accurately identify and delineate BAC regions in the mammograms will be the secondary focus of the outcome assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No